CLINICAL TRIAL: NCT01217281
Title: The Effect of Non-surgical Periodontal Treatment in the Renal Function of Patients With Chronic Kidney Disease: A Randomized Clinical Trial
Brief Title: The Effect of Non-surgical Periodontal Treatment in the Renal Function of Patients With Chronic Kidney Disease: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Spyros Kouris, Spyros Kouris, DIpDS, MClinDent, PhD Candidate, University of Athens
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 143
Record Dates: First submitted 2010-10-06; First posted 2010-10-08 (Estimated); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Chronic Kidney Disease; Periodontitis
Keywords: CKD, Renal, Chronic Kidney Disease, Periodontitis, Perio
MeSH Terms: conditions — Renal Insufficiency, Chronic; Periodontitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Full mouth supra-gingival debridement using hand instruments and ultrasonic scalers, in one session. Patient motivation and oral hygiene instructions Review and prophylaxis at 1 month, 3 months and 6 months after initial treatment session.
  Full mouth periodontal therapy provided at the end of the 6month period (supra and sub- gingival full mouth scaling)
- Test/ Non-surgical Periodontal Therapy (Active Comparator): Full mouth periodontal therapy (sub and supra- gingival debridement) provided under local anaesthesia in two half-mouth sessions.
  Review and prophylaxis 1 month, 3 months and 6 months after the end of the initial therapy.
  Interventions: Procedure: Full Mouth Non-Surgical Periodontal Therapy

INTERVENTIONS:
Procedure: Full Mouth Non-Surgical Periodontal Therapy — Non-surgical Periodontal Therapy provided in two sessions, one for the right half and one for the left half of the dentition. Treatment sessions are provided within one week. No antibiotics or other adjunctive medications are to be used
  Arms: Test/ Non-surgical Periodontal Therapy

SUMMARY:
Periodontal disease is a bacterially-induced inflammation. As such, it can become a point of entry of bacteria, toxins and cytokines into the systemic blood circulation, thus adversely affecting the function of kidneys. This is turn can aggravate the condition of patients with CKD.

The study hypothesis is that periodontal therapy can improve renal function in patients with CKD and lower the blood levels of markers for systemic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Kidney Disease (Stage II, III, IV)
* At least 12 teeth present in the oral cavity
* Moderate to severe chronic periodontitis, which is defined as: at least 8 surfaces with periodontal pocket depth (PPD) ≥5mm and at least 4 surfaces with Clinical Attachment Loss (CAL) ≥4mm, distributed in at least two quadrants.

Exclusion Criteria:

* Patients that have had a renal transplant or undergoing dialysis
* Acute infections or use of antibiotics in the past 3 months.
* Auto-immune diseases, conditions that cause immunosuppression or use of immunosuppressant medication.
* Systemic conditions that require antibiotic prophylaxis for routine periodontal therapy.
* Non-surgical periodontal therapy in the past 6 months or surgical periodontal therapy in the past 12 months.
* Use of medication that can cause gingival hyperplasia such as cyclosporine or fenintoin.
* Myocardial infarction or cerebral vascular incident in the past 12 months or uncontrolled angina.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-01-30 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-06-18 (Actual)

PRIMARY OUTCOMES:
eGFR | 6 months
  Estimated Glomerular Filtration Rate

SECONDARY OUTCOMES:
CRP | 6 months
  C-Reactive Protein level
d-8-iso prostaglandin F2a | 6 months
  d-8-iso prostaglandin F2a
Level of IgG antibodies in serum against periodontal pathogens | 6 months
  Serum samples will be screened for the presence of IgG antibodies against the below mentioned periodontal pathogens, using the "checkerboard immunoblotting" method:
  Porphyromonas gingivalis, Prevotella intermedia, Prevotella nigrescens, Bacteroides forsythus, Treponema denticola, Fusobacterium nucleatum, Actinobacillus actinomycetemcomitans, Campylobacter rectus, Eikenella corrodens, Peptostreptococcus micros, Veillonella parvula, Capnocytophaga ochracea, Streptococcus intermedius, Streptococcus sanguis και Streptococcus oralis.per
Composition of dental plaque | 6 months
  Samples of subgingival plaque will be assessed using DNA probes according to the "checkerboard DNA- DNA hybridization" method. DNA probes will be used against the following bacteria: Porphyromonas gingivalis, Prevotella intermedia, Prevotella nigrescens, Bacteroides forsythus, Treponema denticola, Fusobacterium nucleatum, Actinobacillus actinomycetemcomitans, Campylobacter rectus, Eikenella corrodens, Peptostreptococcus micros, Veillonella parvula, Capnocytophaga ochracea, Streptococcus intermedius, Streptococcus sanguis and Streptococcus oralis
HbA1C | 6 months
  Glycosylated Hemoglobin
FMD / NMD | 6 months
  Flow Mediated Dialation, Nitroglycerin Mediated Dialation, Assessment of Endothelial Dysfunction
PWV | 6 months
  Pass Wave Velocity, Assessment of Endothelial Dysfunction
AIx | 6 months
  Augmentaion Index
Cholesterol levels | 6 months
  Chloesterol Levels
Ca | 6 months
  Serum Calcium
P | 6 months
  Serum Phosphate
Triglycerides | 6 months
  Serum triglycerides
LDL / HDL | 6 months
  Low / High Density Lipoprotein
Serum Urea | 6 months
  Serum Urea
Serum Albumin | 6 months
  Serum Albumin
Urine Albumin | 6 months
  Urine Albumin
Urine Creatinine | 6 months
  Urine Creatinine
Cr/Alb ratio | 6 months
  Urine Creatinine / Albumin Ration

OTHER OUTCOMES:
Periodontal Indices (PPD, CAL, BOP, GI) | 6 months
  Assessment of the periodontal status

CONTACTS AND LOCATIONS:
Overall Officials: Phoebus N Madianos, PhD, Principal Investigator — University of Athens
Locations (1):
- University of Athens, Dental School, Department of Periodontology, Athens, Greece